CLINICAL TRIAL: NCT01818752
Title: A Randomized, Open-label Phase 3 Study of Carfilzomib, Melphalan, and Prednisone Versus Bortezomib, Melphalan, and Prednisone in Transplant-ineligible Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Phase 3 Study of Carfilzomib, Melphalan, Prednisone vs Bortezomib, Melphalan, Prednisone in Newly Diagnosed Multiple Myeloma
Acronym: CLARION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-005; 2012-005283-97 (EudraCT Number); 20130397 (Other: Amgen Inc.)
Record Dates: First submitted 2013-02-12; First posted 2013-03-26 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Bortezomib; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carfilzomib, Melphalan, Prednisone (Experimental): Participants received carfilzomib administered in combination with melphalan and prednisone for nine 42-day cycles. Carfilzomib was administered as an intravenous (IV) infusion on days 1, 2, 8, 9, 22, 23, 29, and 30 of each 42-day cycle. The carfilzomib dose was at 20 mg/m² on cycle 1, days 1 and 2 followed by 36 mg/m² thereafter. On days 1 to 4, melphalan was administered at 9 mg/m² and prednisone was administered at 60 mg/m².
  Interventions: Drug: Carfilzomib; Drug: Melphalan; Drug: Prednisone
- Bortezomib, Melphalan, Prednisone (Active Comparator): Participants received bortezomib in combination with melphalan and prednisone for nine 42-day cycles. Bortezomib was administered either IV or subcutaneously at 1.3 mg/m² during cycles 1 to 4 on days 1, 4, 8, 11, 22, 25, 29, and 32 followed by 1.3 mg/m² during cycles 5 to 9 on days 1, 8, 22, and 29. On days 1 to 4 of each cycle, melphalan was administered at 9 mg/m² and prednisone was administered at 60 mg/m².
  Interventions: Drug: Bortezomib; Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib was administered over 30 minutes on days 1, 2, 8, 9, 22, 23, 29, and 30 for nine 42-day cycles. Carfilzomib 20 mg/m² IV was administered on days 1 and 2 of cycle 1, followed by escalation to 36 mg/m² IV starting on day 8 of cycle 1.
  Other Names: Krypolis®
  Arms: Carfilzomib, Melphalan, Prednisone
Drug: Bortezomib — Bortezomib 1.3 mg/m² was administered as a bolus IV injection or as a subcutaneous injection (per investigator's choice, dose modification, or regulatory approval) on days 1, 4, 8, 11, 22, 25, 29, and 32 of cycles 1 to 4, and on days 1, 8, 22, and 29 of cycles 5 to 9.
  Other Names: Velcade®
  Arms: Bortezomib, Melphalan, Prednisone
Drug: Melphalan — Melphalan 9 mg/m² was taken orally on days 1 to 4 of all cycles.
Drug: Prednisone — Prednisone 60 mg/m² was taken orally on days 1 to 4 of all cycles.

SUMMARY:
The primary objective was to compare the progression-free survival of transplant ineligible patients newly diagnosed with multiple myeloma who were treated with carfilzomib, melphalan and prednisone (CMP) or with Velcade® (bortezomib), melphalan and prednisone (VMP).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed symptomatic multiple myeloma (per International Myeloma Working Group [IMWG] diagnostic criteria)
2. Transplant ineligibility
3. Measurable disease, as defined by 1 or more of the following (assessed within 21 days prior to randomization):

   * Serum M-protein ≥ 0.5 g/dL, or
   * Urine M-protein ≥ 200 mg/24 hours, or
   * In subjects without detectable serum or urine M-protein, serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal kappa lambda ratio (SFLC kappa lambda ratio < 0.26 or > 1.65)
4. No prior treatment for multiple myeloma
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

1. Multiple myeloma of IgM (immunoglobulin M) subtype
2. Glucocorticoid therapy within 14 days prior to randomization that equals or exceeds a cumulative dose of 160 mg of dexamethasone
3. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
4. Plasma cell leukemia (> 2.0 × 10^9/L circulating plasma cells by standard differential)
5. Waldenström macroglobulinemia (WM)
6. Known amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 955 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (212):
- United States (14):
  - California Cancer Associates for Research & Excellence, Inc. (cCARE), Fresno, California
  - Marin Cancer Care, Greenbrae, California
  - Sutter Gould Medical Foundation, Modesto, California
  - Innovative Clinical Research Institute, Whittier, California
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - Evanston KelIogg Cancer Center, Evanston, Illinois
  - Billings Clinic Cancer Center, Billings, Montana
  - Maimonides Cancer Center, Brooklyn, New York
  - Weill Cornell Medical Center, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Saint Francis Health System, Greenville, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Santee Hematology Oncology, Sumter, South Carolina
  - Seattle Cancer Care Alliance, Seattle, Washington
- Argentina (2):
  - Centro de educacion medica c investigacioncs clinicas "Norberto Quimo' (CEMIC), Buenos Aires
  - Sanatorio Britanico S.A., Santa Fe
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Central Coast Local Health District, North Gosford, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Royal North Shore Hospital, Haematology Department, New South Wales
- Austria (3):
  - Medical University of Innsbruck, University Clinic for Internal Medicine V, Innsbruck
  - Elisabeth Linz Hospital, Linz
  - Vienna Wilhelminen Hospital, Vienna
- Belgium (4):
  - ZNA, Stuivenberg, Antwerp, Antwerpen
  - Saint Joseph Clinic Arlon, Department of Hematology, Arlon, Luxembourg
  - CHR de La Citadelle (ENG: Citadelle Regional Hospital Center), Liège
  - CHU Mont-Godinne, Yvoir
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Hematology Clinic, Plovdiv
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Oncology and Hematology Clinic, Plovdiv
  - Military Medical Academy - Multiprofile Hospital for Active Treatment, Sofia, Hematology and Oncology Clinic, Sofia
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia, Hematology Clinic, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna, Varna
- CSSS-Champlain-Charles LeMoyne, Greenfield Park, Quebec, Canada
- China (16):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of the Fourth Military Medical University of PLA, Xi’an, Shanxi
  - The First Affiliated Hospital of College of Medicine, Zhejiang University - Dr. Jie Jin, Hangzhou, Zhejiang
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - 307 Hospital of PLA, Beijing
  - Beijing Chao Yang Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Institute on Hematology & Blood Diseases Hospital Chinese Academy of Medical Scicnces & Peking Union Medical University, Tianjin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
- Czechia (7):
  - University Hospital Brno, Department of Internal Hematology and Oncology, Brno
  - University Hospital Brno, Hospital Pharmacy - Department of Dilution of Cytostasis, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, 3rd Clinic of Internal Medicine, Nephrology, Rheumatology and Endocrinology, Olomouc
  - University Hospital Ostrava, Clinic of Hematooncology of UHO and MFUO, Ostrava
  - University Hospital Kralovske Vinohrady - Internal Hematology Clinic, Prague
  - General University Hospital Prague, 1st Department of Medicine - Department of Hematology, Prague
- France (16):
  - CHU de Caen, Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - UHC Dijon, Children's Hospital, Dijon
  - CHRU Lille Hôpital Claude Huriez, Lille
  - CHRU Hopital Huriez, Departement of Hematology, Lille
  - Paoli Calmettes Institute, Department ofHematology 2, Marseille
  - Nantes University Hospital Center, Nantes
  - Centre Hospitalier Regional Universitaire de Nimes, Groupe Hospitalo-Universitaire Caremeau, Nîmes
  - Hopital Saini Louis, Service d'immuno-Hematologie, Paris
  - Hopital Saint Antoine, Paris
  - Hospital Necker, Paris
  - South Lyon Hospital Center, Pierre-Bénite
  - Centre Hospitalier Lyon Sud, Service d'hématologie Clinique, Pierre-Bénite
  - Hopital Pontchaillou, Rennes
  - Hospital Purpan, Toulouse
  - CHU de Tours Hopital Bretonneau, Tours
- Germany (8):
  - Freiburg University Medical Center, Freiburg im Breisgau, Baden-Wurttemberg
  - Ulm University Hospital, Center for Internal Medicine, Clinic of Internal Medicine III, Ulm, Baden-Wurttemberg
  - Ludwig Maximilians University Hospital - Medical Clinic III, Munich, Bavaria
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - Johannes Gutenberg-University Mainz, Medical Clinic and Policlinic III, Mainz, Rhineland-Palatinate
  - Saarland University Hospital, Homburg / Saar, Saarland
  - Group Practice for Hematology and Oncology, Dresden
  - Stiftungsklinikum Mittelrhein GmbH, Clinic of Internal Medicine, Koblenz
- Greece (2):
  - Evangelismos Hospital, Athens, Attica
  - University of Athens, Alexandra Hospital, Athens
- Hungary (7):
  - St. Istvan and St. Laszlo Hospital of Budapest, Department of Haematology and Stem-cell Transplant, Budapest
  - National Institute of Oncology, Department of Oncology, Internal Medicine "A" and Hematology, Budapest
  - University of Debrecen, Medical and Health Science Center, Institute for Medicine, Chair of Hematology, Debrecen
  - Bekes County Pandy Kalman Hospital 1st Department of Internal Medicine, Hematology, Gyula
  - Kaposi Mor County Teaching Hospital, 2nd Department of Internal Medicine, Hematology, Kaposvár
  - Bacs-Kiskun County Teaching Hospital, II. Department of Internal Medicine, Kecskemét
  - Medical Center of the University of Pecs, 1st Clinic for Internal Medicine, Pécs
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Department of Hematology, Haifa
  - Ein Kerem Hospital, Department of Hematology, Jerusalem
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (8):
  - UO Clinica Ematologica, IRCCS A.O.U. San Martino, Genova, GE
  - A.O.U. San Luigi Gonzaga, Orbassano, TO
  - Ospedali Riuniti di Ancona Umberto I, G.M. Lancisi, G. Salesi, Ancona
  - Maggiore della Carita Hospital of Novara, Novara
  - Local NHS of Piacenza Hospital Guglielmo da Saliceto Department Oncology-Hematology, Unit of Hema, Piacenza
  - Ospedale S. Eugenio, Roma
  - Policlinico Universitario "Umberto I", Rome
  - AO Città della Salute e della Scienza di Torino, Division of Hematology, Torino
- Japan (16):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - National Hospitalization Organization Kyushu Cancer Center, Minamiku, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Osaka University Hospital, Suita, Osaka
  - Japanese Red Cross Medical Center, Tokyo, Shibuya-ku
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Koto, Tokyo
  - National Center for Global Health and Medicine, Shinjuku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Tokushima Prefectural Central Hospital, Tokushima
- Mexico (4):
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Fundacion Centro Oncologieo de Integracion Regional - COIR, Mendoza
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Consultorio Privado del Dr. Guillermo Jose Ruiz y Arguelles, Puebla City
- Netherlands (4):
  - Vrije Universiteit Medisch Centrum (VUMC), Department of Hematology, Amsterdam
  - St. Antonius Ziekenhuis, Department of Hematology, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - Isala Clinics in Zwolle, Department of Oncology, Zwolle
- New Zealand (4):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - Canterbury Health Laboratories, Christchurch
  - Wellington Hospital, Wellington
- Poland (8):
  - Independent Public Healthcare Facility of the Ministry of Internal Affairs & Warminsko-Mazurskie Oncology Centre in Olsztyn, Olsztyn, OIsztyn
  - Independent Public Healthcare Facility Municipal Hospital Group, Department of Hematology, Chorzów, Silesian Voivodeship
  - Andrzej Mielecki Independent Public Clinical Hospital of Medical University of Silesia in Katowice, Katowice
  - Independent Public Healthcare Facility University Hospital, Krakow
  - Nicolaus Copernicus Memorial Provincial Specialist Hospital, Lodz
  - Independent Public Teaching Hospital No.1 in Lublin, Dept. of Hematology-Oncology, Lublin
  - Nicolaus Copernicus Municipal Specialist Hospital, Department of Hematology, Torun
  - Maria Sklodowska-Curie Institute of Oncology, Warsaw
- Romania (7):
  - "Prof. Dr. Ion Chiricuta" Institut of Oncology, Hematology Department, Cluj-Napoca, Cluj
  - Iasi Regional Institute for Oncology, Medical Hematology Department, Iași, Iaşi
  - Brasov County Emergency Clinical Hospital, Hematology Department, Brasov
  - Fundeni Clinical Institute, Hematology Department, Bucharest
  - Coltea Clinical Hospital, Hematology Department, Bucharest
  - Bucharest Emergency University Hospital, Hematology Department, Bucharest
  - Targu-Mures County Emergency Clinical Hospital, Clinic of Hematology and Bone Marrow Transplantation, Târgu Mureş
- Russia (9):
  - State Medical Institution: Republican Hospital n a.V.A. Baranov, Department of Hematology, Petrozavodsk, Republic of Karelia
  - Arkhangelsk Regional Clinical Hospital, Department of internal diseases #2, Arkhangelsk
  - State Medical Institution: First Republican Clinical Hospital under the Ministry of Healthcare of the Republic of Udmurtia, Izhevsk
  - Institution of the Russian Academy of Medical Sciences Russian Oncological Research Center n.a. N.N.Blokhin under the Russian Academy of Medical Sciences, Moscow
  - City Clinical Hospital N.A.S.P. Botkin, Department of Bone Marrow Transplantation and Intensive Chemotherapy for Patients with Myeloproliferative Disorders, Moscow
  - Federal State Institution: Russian Research Institute of Hematology and Blood Transfusion under the Federal Agency for High-Tech Medical Care, Saint Petersburg
  - City Clinical Hospital #31, Department of Bone Marrow Transplantation and Intensive Chemotherapy for Patients with Myeloproliferative Disorders, Saint Petersburg
  - State Higher Educational Institution St. Petersburg Pavlov State Medical University, Saint Petersburg
  - The Federal State Budget Institute The Nikiforov Russian Center of Emergency and Radiation Medicine the Ministry of Russian, Saint Petersburg
- Singapore (4):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Singapore Oncology Consultants, Gleneagles Hospital, Singapore
  - OncoCare Cancer Center, Singapore
- South Korea (12):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Pusan National University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barselona
  - University Hospital of Navarra, Pamplona, Navarre
  - Hospital Clinic i Provincial Barcelona, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario, Salamanca, Salamanca
  - Hospital Virgen del Rocio University, Seville
  - Universitari i Politècnic la Fe de Valencia Consulta Externa de Hematología, Valencia
  - Hospital Quiron Zaragoza, Zaragoza
- Switzerland (2):
  - University Hospital Center Vaudois, Lausanne
  - County Hospital Saint Gallen, Sankt Gallen
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Kuohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Linkou, Tapei
- Turkey (Türkiye) (3):
  - Ege University Medical Faculty, Izmir, Bornova
  - Ankara University Medical Faculty, Cebeci Research and Application Hospital, Hematology Department, Ankara, Cebeci
  - Marmara University Pendik Training and Research Hospital, Istanbul, Pendik
- Ukraine (10):
  - Cherkasy Regional Oncology Center, Cherkasy
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Hematology Centre, Dnipropetrovsk
  - Kharkiv Regional Clinical Oncology Center, Department of Hematology, Kharkiv
  - Khmelnytskyi Regional Hospital, Hematology Department, Khmelnytskyi
  - Kyiv Center for Bone Marrow Transplantation, Kyiv
  - Institute of Blood Pathology and Transfusion Medicine, Lviv
  - Poltava M.V. Sklifosovskyi Regional Clinical-Hospital, Poltava
  - A. Novak Zakarpattia Regional Clinical Hospital, Uzhhorod
  - M.I. Pyrohov Vinnytsya Regional Clinical Hospital, Hematology Department, Vinnitsya
  - O.F. Herbachevskyi Regional Clinical Hospital, Hematology Center, Zhytomyr
- United Kingdom (8):
  - Kent and Canterbury Hospital, Canterbury, Kent
  - Maidstone Hospital, Kent Oncology Centre, Maidstone, Kent
  - Northwick Park Hospital, Harrow, Middlesex
  - Raigmore Hospital, Inverness
  - University College London, Cancer Centre, London
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - Oxford University Hospitals NHS Trust, Churchill Hospital, Oxford
  - The Royal Wolverhampton Hospitals NHS Trust, New Cross Hospital, Wolverhampton

REFERENCES:
- [Background] Chari A, Stewart AK, Russell SD, Moreau P, Herrmann J, Banchs J, Hajek R, Groarke J, Lyon AR, Batty GN, Ro S, Huang M, Iskander KS, Lenihan D. Analysis of carfilzomib cardiovascular safety profile across relapsed and/or refractory multiple myeloma clinical trials. Blood Adv. 2018 Jul 10;2(13):1633-1644. doi: 10.1182/bloodadvances.2017015545. PMID 29991494
- [Background] Facon T, Lee JH, Moreau P, Niesvizky R, Dimopoulos M, Hajek R, Pour L, Jurczyszyn A, Qiu L, Klippel Z, Zahlten-Kumeli A, Osman M, Paiva B, San-Miguel J. Carfilzomib or bortezomib with melphalan-prednisone for transplant-ineligible patients with newly diagnosed multiple myeloma. Blood. 2019 May 2;133(18):1953-1963. doi: 10.1182/blood-2018-09-874396. Epub 2019 Feb 28. PMID 30819926
- [Derived] Rosenthal A, Luthi J, Belohlavek M, Kortum KM, Mookadam F, Mayo A, Fonseca R, Bergsagel PL, Reeder CB, Mikhael JR, Stewart AK. Carfilzomib and the cardiorenal system in myeloma: an endothelial effect? Blood Cancer J. 2016 Jan 15;6(1):e384. doi: 10.1038/bcj.2015.112. PMID 26771810
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 183 centers in Argentina, Australia, Austria, Belgium, Bulgaria, Canada, China, Czech Republic, France, Germany, Greece, Hungary, Israel, Italy, Japan, Mexico, Netherlands, New Zealand, Poland, Romania, Russia, Singapore, South Korea, Spain, Switzerland, Taiwan, Turkey, Ukraine, United Kingdom, and United States.
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio. Randomization was stratified by International Staging System (ISS) stage (stage 1 versus stages 2 or 3), choice of route of bortezomib administration (intravenous [IV] versus subcutaneous [SC]), region (North America, Europe, Asia Pacific, or other), and age (< 75 years versus ≥ 75 years).
Period: Overall Study
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Started | 477 | 478
Received Treatment | 470 | 474
Completed | 290 (Completed treatment) | 280 (Completed treatment)
Not Completed | 187 | 198
Not completed — Adverse Event | 64 | 74
Not completed — Death | 14 | 18
Not completed — Non-compliance | 16 | 20
Not completed — Withdrawal by Subject | 15 | 14
Not completed — Physician Decision | 9 | 8
Not completed — Disease Progression | 54 | 48
Not completed — Other | 7 | 8
Not completed — Continuing Treatment | 1 | 4
Not completed — Randomized but not Dosed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone | Total
Number analyzed (Participants) | 477 | 478 | 955
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (6.5) | 72.0 (5.7) | 71.7 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 235 | 473
  Male | 239 | 243 | 482
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 33
  Not Hispanic or Latino | 443 | 427 | 870
  Unknown or Not Reported | 19 | 33 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 121 | 123 | 244
  Black or African American | 0 | 3 | 3
  White | 339 | 329 | 668
  Other | 3 | 1 | 4
  Multiple | 0 | 2 | 2
  Not Reported | 12 | 19 | 31
Stratification Factor: International Staging System (ISS) Stage [Number; unit: participants] — The International Staging System (ISS) for myeloma was published by the International Myeloma Working Group:
  * Stage I: β2-microglobulin (β2M) < 3.5 mg/L, albumin >= 3.5 g/dL
  * Stage II: β2M < 3.5 mg/L and albumin < 3.5 g/dL; or β2M 3.5 mg/L - 5.5 mg/L irrespective of the serum albumin
  * Stage III: β2M ≥ 5.5 mg/L
  participants
    Stage I | 99 | 95 | 194
    Stage II or III | 378 | 383 | 761
Stratification Factor: Route of Bortezomib Administration [Number; unit: participants] — The route of bortezomib administration (IV versus SC) was made per investigator's choice, dose modification, or regulatory approval. The investigator selected the route for all participants prior to randomization to treatment group in order to minimize any evaluation bias because of imbalances in potential prognostic factors that might have impacted the investigator's choice of a particular route.
  participants
    Intravenous | 123 | 123 | 246
    Subcutaneous | 354 | 355 | 709
Stratification Factor: Region of Enrollment [Number; unit: participants]
  Asia Pacific | 141 | 140 | 281
  North America | 12 | 8 | 20
  Europe | 317 | 320 | 637
  Other | 7 | 10 | 17
Stratification Factor: Age [Number; unit: participants]
  < 75 years | 329 | 327 | 656
  ≥ 75 years | 148 | 151 | 299
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Dead.
  participants
    0 (Fully active) | 125 | 129 | 254
    1 (Restrictive but ambulatory) | 250 | 260 | 510
    2 (Ambulatory but unable to work) | 101 | 89 | 190
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to the earlier of documented disease progression or death due to any cause. PFS was analyzed using Kaplan-Meier methods. The duration of PFS was censored for participants with no baseline and/or post-baseline disease assessments, who started a new anti-cancer therapy before documentation of disease progression or death, death or disease progression after missed disease assessment of 100 consecutive days or longer, or who were alive without documentation of disease progression before the data cutoff date, including lost to follow-up prior to disease progression.
  Participants were evaluated for disease response and progression according to the International Myeloma Working Group Uniform Response Criteria (IMWG-URC), determined centrally using a validated computer algorithm in a blinded manner.
Time Frame: From randomization until the data cut-off date of 15 July 2016; median follow-up time for PFS was 21.6.and 22.2 months in the bortezomib and carfilzomib arms respectively.
Population: The intent-to-treat population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Number analyzed (Participants) | 477 | 478
months | 22.1 [20.8 to 24.4] | 22.3 [20.9 to 26.7]
Statistical Analysis 1: Comparison: Bortezomib, Melphalan, Prednisone vs Carfilzomib, Melphalan, Prednisone; The inferential test associated with the primary analysis of PFS was assessed against an overall 1-sided significance level of α=0.025; Test type: Superiority or Other; p = 0.1590, Log Rank — The p-value boundary for PFS analysis was 0.02141; Log-rank p-value (1-sided) stratified by ISS stage, choice of route of bortezomib administration, region and age; Hazard Ratio (HR) = 0.906, 95% CI 2-sided [0.746 to 1.101] — The hazard ratio (Carfilzomib/Bortezomib) was estimated using a Cox proportional hazards model stratified by ISS stage, choice of route of bortezomib administration, region and age

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from randomization to the date of death (whatever the cause). Participants who were alive or lost to follow-up as of the data analysis cut-off date were censored on the date the patient was last known to be alive.
  Median overall survival was estimated using the Kaplan-Meier method.
Time Frame: From randomization until the data cut-off date of 15 July 2016; median follow-up time for OS was 22.2 and 22.5 months in the bortezomib and carfilzomib arms respectively.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Number analyzed (Participants) | 477 | 478
months | NA [NA to NA] — Not estimable due to the low number of events | NA [31.5 to NA] — Not estimable due to the low number of events
Statistical Analysis 1: Comparison: Bortezomib, Melphalan, Prednisone vs Carfilzomib, Melphalan, Prednisone; Test type: Superiority or Other; p = 0.8934, Log Rank — Based on the pre-specified multiplicity adjustment method, secondary endpoints were to be tested only if the results of the primary endpoint were significant. The p-values for all secondary endpoints are descriptive only; Log-rank p-value (1-sided) stratified by ISS stage, choice of route of bortezomib administration, region and age; Hazard Ratio (HR) = 1.211, 95% CI 2-sided [0.896 to 1.637] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response Rate
Description: Disease response was evaluated according to the IMWG-URC using a validated computer algorithm. Overall response was defined as the percentage of participants with a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
  sCR: As for CR, normal serum free light chain (SFLC) ratio and no clonal cells in bone marrow (BM).
  CR: No immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and < 5% plasma cells in BM biopsy; VGPR: Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% reduction in serum M-protein with urine M-protein <100 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
  PR: ≥ 50% reduction of serum M-protein and reduction in urine M-protein by ≥ 90% or to < 200 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
Time Frame: Disease response was assessed every 3 weeks during the first 54 weeks and every 6 weeks thereafter until PD or the data cut-off date of 15 July 2016; median follow-up time was 21.6.and 22.2 months in the bortezomib and carfilzomib arms respectively.
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Number analyzed (Participants) | 477 | 478
percentage of participants | 78.8 [74.9 to 82.4] | 84.3 [80.7 to 87.5]
Statistical Analysis 1: Comparison: Bortezomib, Melphalan, Prednisone vs Carfilzomib, Melphalan, Prednisone; Test type: Superiority or Other; p = 0.0218, Stratified Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Cochran-Mantel-Haenszel Chi-square test stratified by ISS stage, choice of route of bortezomib administration, region and age; Odds Ratio (OR) = 1.412, 95% CI 2-sided [1.010 to 1.973] — Odds ratio (Carfilzomib/Bortezomib) was estimated using the Mantel-Haenszel method stratified by ISS stage, choice of route of bortezomib administration, region and age

4. Secondary Outcome: Complete Response Rate
Description: Complete response rate was defined as the percentage of participants in each treatment group who achieved a sCR or CR per the IMWG-URC as their best response.
  sCR: As for CR, normal serum free light chain (SFLC) ratio and no clonal cells in bone marrow (BM).
  CR: No immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and < 5% plasma cells in BM biopsy.
Time Frame: as for outcome 3
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Number analyzed (Participants) | 477 | 478
percentage of participants | 23.1 [19.4 to 27.1] | 25.9 [22.1 to 30.1]
Statistical Analysis 1: Comparison: Bortezomib, Melphalan, Prednisone vs Carfilzomib, Melphalan, Prednisone; Test type: Superiority or Other; p = 0.1388, Stratified Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.179, 95% CI 2-sided [0.875 to 1.589] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants With ≥ Grade 2 Peripheral Neuropathy
Description: Neuropathy events were defined as Grade 2 or higher peripheral neuropathy as specified by peripheral neuropathy Standardised Medical Dictionary for Regulatory Activities (MedDRA) Query, narrow (scope) (SMQN) terms.
  Peripheral neuropathy was assessed by neurologic exam and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03:
  Grade 1: Asymptomatic; Grade 2: Moderate symptoms, limiting instrumental activities of daily living (ADL) Grade 3: Severe symptoms; limiting self-care ADL; Grade 4: Life-threatening consequences, urgent intervention indicated; Grade 5: Death.
Time Frame: From the first dose of any study drug up to 30 days after the last dose of any study drug as of the data cut-off date of 15 July 2016; median duration of treatment was 52 weeks in both treatment groups.
Population: The safety population included all randomized participants who received at least 1 dose of any study treatment (i.e., carfilzomib, bortezomib, melphalan, or prednisone).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Number analyzed (Participants) | 470 | 474
percentage of participants | 35.1 [30.8 to 39.6] | 2.5 [1.3 to 4.4]
Statistical Analysis 1: Comparison: Bortezomib, Melphalan, Prednisone vs Carfilzomib, Melphalan, Prednisone; Test type: Superiority or Other; p < 0.0001, Pearson Chi-Square test — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.048, 95% CI 2-sided [0.026 to 0.088] — Unstratified odds ratio (Carfilzomib/Bortezomib) was estimated

6. Secondary Outcome: European Organisation for Research and Treatment of Cancer Quality of Life Core Module (EORTC QLQ-C30) Global Health Status/Quality of Life (QOL) Scores
Description: The EORTC QLQ-C30 is a validated self-rating questionnaire including 30 items used to assess the overall quality of life in cancer patients.
  It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact).
  The EORTC QLQ-C30 Global Health Status/QOL scale was scored between 0 and 100, with higher scores indicating better Global Health Status/QOL.
Time Frame: Baseline, weeks 6, 12, 18, 24, 30, 36, 42 and 48
Population: Intent-to treat population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Number analyzed (Participants) | 477 | 478
units on a scale
  Baseline (n = 425, 425) | 53.3 (21.9) | 53.9 (22.5)
  Week 6 (n = 412, 407) | 56.2 (19.5) | 61.1 (19.6)
  Week 12 (n = 376, 389) | 55.3 (19.8) | 62.4 (17.7)
  Week 18 (n = 341, 369) | 55.7 (18.8) | 63.2 (17.4)
  Week 24 (n = 320, 345) | 57.3 (17.6) | 63.3 (17.1)
  Week 30 (n = 298, 317) | 61.6 (17.8) | 63.0 (17.8)
  Week 36 (n = 285, 308) | 61.9 (17.5) | 64.0 (18.1)
  Week 42 (n = 275, 288) | 63.3 (17.7) | 65.0 (18.1)
  Week 48 (n = 261, 265) | 62.9 (18.4) | 65.1 (17.1)
Statistical Analysis 1: Comparison: Bortezomib, Melphalan, Prednisone vs Carfilzomib, Melphalan, Prednisone; Treatment groups were compared using a linear mixed model for repeated measures (MMRM). The model included the fixed, categorical effects of treatment (all baseline responses were modeled with a dummy treatment), the randomization stratification factors - ISS stage, choice of route of bortezomib administration, region, age, and random effects of subject intercept and coefficient on time; Test type: Superiority or Other; p < 0.0001, Mixed Effects Model for Repeated Measure — [p-value comment as in outcome 2, analysis 1]; Least squares mean difference = 4.99, 95% CI 2-sided [3.48 to 6.51], Standard Error of Mean 0.773

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs)were graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.03, where GRADE 1 = Mild; GRADE 2 = Moderate; GRADE 3 = Severe; GRADE 4 = Life-threatening; GRADE 5 = Fatal.
  A serious adverse event is an adverse event that met 1 or more of the following criteria:
  * Death
  * Life-threatening
  * Required inpatient hospitalization or prolongation of an existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Congenital anomaly/birth defect
  * Important medical event that jeopardized the participant and may have required medical or surgical intervention to prevent 1 of the outcomes listed above.
  Treatment-related adverse events are adverse events considered related to at least 1 investigational product by the investigator, including those with unknown relationship.
Time Frame: as for outcome 5
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Number analyzed (Participants) | 470 | 474
participants
  All adverse events | 454 | 460
  AEs ≥ grade 3 | 358 | 354
  Serious adverse events | 198 | 235
  Leading to discontinuation of study drug | 73 | 83
  Fatal adverse events | 20 | 31
  Treatment-related adverse events (TRAEs) | 431 | 408
  TRAEs ≥ grade 3 | 285 | 268
  Treatment-related serious adverse events | 102 | 136
  TRAE leading to discontinuation of study drug | 51 | 54
  Treatment-related fatal adverse events | 5 | 10

ADVERSE EVENTS:
Time Frame: From the first dose of any study drug up to 30 days after the last dose of any study drug as of the data cut-off date of 15 July 2016; median duration of treatment was 52 weeks in both treatment groups.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Bortezomib, Melphalan, Prednisone | Carfilzomib, Melphalan, Prednisone
Serious Adverse Events (participants affected / at risk) | 198/470 | 235/474
Other Adverse Events (participants affected / at risk) | 437/470 | 437/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib, Melphalan, Prednisone (N=470) | Carfilzomib, Melphalan, Prednisone (N=474)
Anaemia (Blood and lymphatic system disorders) | 6 | 11
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 4
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 5
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 4
Angina pectoris (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 7
Atrial flutter (Cardiac disorders) | 1 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac amyloidosis (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 7 | 21
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 8
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Hypertensive cardiomegaly (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 | 0
Diplopia (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 5 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 6 | 4
Chest pain (General disorders) | 1 | 2
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 5 | 2
Generalised oedema (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1
Infusion site pain (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 9 | 16
Sudden death (General disorders) | 1 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 3 | 8
Cellulitis (Infections and infestations) | 0 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 2
Hepatitis C (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 3
Influenza (Infections and infestations) | 0 | 2
Legionella infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 6 | 5
Otitis media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 31 | 46
Postoperative wound infection (Infections and infestations) | 0 | 1
Pseudomonas bronchitis (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 7 | 8
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 3 | 5
Urosepsis (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 4
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Heat illness (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 2
Blood uric acid increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 3 | 2
Urine output decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Tetany (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Autonomic neuropathy (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Coma (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Hypotonia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 5 | 4
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 3
Hallucination (Psychiatric disorders) | 1 | 0
Illusion (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 10 | 19
Chronic kidney disease (Renal and urinary disorders) | 1 | 3
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 14
Renal impairment (Renal and urinary disorders) | 1 | 1
Renal injury (Renal and urinary disorders) | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Immobile (Social circumstances) | 1 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 1 | 0
Bone operation (Surgical and medical procedures) | 1 | 0
Vertebroplasty (Surgical and medical procedures) | 0 | 2
Aortic dissection (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 8
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 7 | 3
Hypovolaemic shock (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib, Melphalan, Prednisone (N=470) | Carfilzomib, Melphalan, Prednisone (N=474)
Anaemia (Blood and lymphatic system disorders) | 143 | 168
Leukopenia (Blood and lymphatic system disorders) | 39 | 34
Neutropenia (Blood and lymphatic system disorders) | 121 | 121
Thrombocytopenia (Blood and lymphatic system disorders) | 91 | 84
Abdominal distension (Gastrointestinal disorders) | 27 | 10
Abdominal pain (Gastrointestinal disorders) | 27 | 12
Abdominal pain upper (Gastrointestinal disorders) | 32 | 21
Constipation (Gastrointestinal disorders) | 114 | 65
Diarrhoea (Gastrointestinal disorders) | 132 | 95
Nausea (Gastrointestinal disorders) | 132 | 167
Vomiting (Gastrointestinal disorders) | 88 | 116
Asthenia (General disorders) | 67 | 70
Chest pain (General disorders) | 11 | 24
Chills (General disorders) | 14 | 44
Fatigue (General disorders) | 85 | 78
Oedema peripheral (General disorders) | 54 | 84
Pyrexia (General disorders) | 80 | 168
Bronchitis (Infections and infestations) | 39 | 40
Nasopharyngitis (Infections and infestations) | 33 | 31
Pneumonia (Infections and infestations) | 27 | 30
Upper respiratory tract infection (Infections and infestations) | 50 | 49
Urinary tract infection (Infections and infestations) | 26 | 29
Alanine aminotransferase increased (Investigations) | 16 | 28
Blood creatinine increased (Investigations) | 22 | 35
Neutrophil count decreased (Investigations) | 71 | 55
Platelet count decreased (Investigations) | 61 | 48
Weight decreased (Investigations) | 24 | 15
White blood cell count decreased (Investigations) | 58 | 51
Decreased appetite (Metabolism and nutrition disorders) | 88 | 67
Hyperglycaemia (Metabolism and nutrition disorders) | 37 | 30
Hyperuricaemia (Metabolism and nutrition disorders) | 22 | 28
Hypocalcaemia (Metabolism and nutrition disorders) | 41 | 47
Hypokalaemia (Metabolism and nutrition disorders) | 63 | 53
Hyponatraemia (Metabolism and nutrition disorders) | 24 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 56 | 53
Bone pain (Musculoskeletal and connective tissue disorders) | 29 | 31
Pain in extremity (Musculoskeletal and connective tissue disorders) | 46 | 30
Dizziness (Nervous system disorders) | 39 | 45
Headache (Nervous system disorders) | 23 | 44
Hypoaesthesia (Nervous system disorders) | 26 | 14
Neuralgia (Nervous system disorders) | 45 | 2
Neuropathy peripheral (Nervous system disorders) | 154 | 29
Paraesthesia (Nervous system disorders) | 32 | 24
Peripheral sensory neuropathy (Nervous system disorders) | 64 | 8
Polyneuropathy (Nervous system disorders) | 36 | 5
Insomnia (Psychiatric disorders) | 65 | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 63
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 72
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 41
Rash (Skin and subcutaneous tissue disorders) | 47 | 26
Hypertension (Vascular disorders) | 32 | 102
Hypotension (Vascular disorders) | 37 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.